CLINICAL TRIAL: NCT00628303
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Trial of the Effect of Motavizumab Prophylaxis on Reduction of the Incidence of Serious Early Childhood Wheezing in Preterm Infants
Brief Title: A Phase 3 Trial of the Effect of Motavizumab Prophylaxis on Reduction of Serious Early Childhood Wheezing in Infants
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study never officially opened for enrollment
Sponsor: MedImmune LLC (Industry)
Responsible Party: Hasan S. Jafri, M.D., MedImmune Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP169
Record Dates: First submitted 2008-02-20; First posted 2008-03-05 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Wheezing
Keywords: Good health
MeSH Terms: conditions — Respiratory Sounds | interventions — motavizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Motavizumab
  Interventions: Biological: Motavizumab
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Motavizumab — 15 mg/kg administered by IM injection every 30 days during the RSV season for a total of 5-6 injections
  Other Names: MEDI-524
  Arms: 1
Other: Placebo — 15 mg/kg administered by IM injection every 30 days during the RSV season for a total of 5-6 injections
  Arms: 2

SUMMARY:
The primary objective of this study is to assess the efficacy of motavizumab compared to placebo when administered monthly to preterm infants during their first RSV season for the reduction of the incidence of serious early childhood wheezing from their 2nd through 3rd birthdays.

DETAILED DESCRIPTION:
The primary objective of this study is assess the efficacy of motavizumab compared to placebo when administered monthly by intramuscular (IM) injection during the first RSV season for the reduction of the incidence of serious early childhood wheezing in preterm infants between their 2nd and 3rd birthdays.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infants born at 32 & 1/7 - 35 & 0/7 weeks GA, determined according to available medical records
* Chronological age of <6 months of age at randomization
* In good health, in the opinion of the investigator
* Not more than one of the following AAP-defined risk factors:

  1. Childcare attendance
  2. School-aged siblings
  3. Exposure to environmental air pollutants (not including passive exposure to tobacco smoke)
* Ability and willingness of the subject's parent/legal guardian to complete all protocol-mandated follow-up telephone contacts, visits and procedures
* Written informed consent obtained from the subject's parent(s) or legal guardian

Exclusion Criteria:

* Diagnosis of CLD of prematurity (also referred to as BPD) or other chronic pulmonary diseases
* Diagnosis of hemodynamically significant CHD, defined as requiring medication or supplemental oxygen for their CHD
* Congenital abnormalities of the airways
* Severe neuromuscular disease, as determined by the investigator
* Previous or concurrent treatment with palivizumab or intravenous immunoglobulin (IVIG)
* Eligible for prophylaxis based on local medical standards and guidelines at participating sites
* Known immunodeficiency
* Previous or current diagnosis of an upper or lower respiratory infection by a medical professional
* Previous or current diagnosis of wheezing, asthma, or other wheezing-related diagnoses
* Hospitalization at the time of enrollment (in case admitted to nursery as part of routine care, infant should only be randomized immediately prior to being discharged)
* Any illness or condition that would preclude long-term survival
* Participation in a trial or an investigational agent for RSV prophylaxis or therapy
* Inability to be followed through their 3rd birthday

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of serious early childhood wheezing episodes | Between 2nd and 3rd birthdays

SECONDARY OUTCOMES:
Frequency of medically-attended lower respiratory tract wheezing events | During 2nd and 3rd birthday
Frequency of medically-attended lower respiratory tract wheezing events from randomization through 3 years of age | From randomization through 3 yrs.
Incidence of serious RSV disease | Through Day 150